CLINICAL TRIAL: NCT03580408
Title: A Prospective Phase II Study Of Nivolumab Alone, Or In Combination With Vinblastin In Patients Aged 61 Years And Older, With Classical Hodgkin Lymphoma And Coexisting Medical Conditions.
Brief Title: Study Of Nivolumab Alone, Or In Combination With Vinblastin In Patients With Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIVINIHO
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Hodgkin Lymphoma; Coexisting Medical Conditions
Keywords: Nivolumab; Lymphoma; Anti-PD1
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Nivolumab; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Induction treatment :Nivolumab will be given alone at 240 mg flat dose every 2 weeks (i.e. one cycle) Patients will be assessed after 3 months of therapy (after 6 injections of Nivolumab)
  Consolidation treatment:
  It depends on the induction evaluation by PET-CT and CT-scan (Lugano 2014 criteria) :
  * For patients achieving CMR according to Lugano Classification : treatment by nivolumab 240 mg every 2 weeks for 9 months.
  * Patients who reach PMR and NMR after 3 months (according to Lugano Classification) will be treated by the Nivolumab+Vinblastin regimen every 2 weeks for 9 additional months: Vinblastin(6 mg/m2 (IV) + Nivolumab 240 mg (IV)
  * In case of progressive disease , patients will be considered in treatment failure.
  Interventions: Drug: Nivolumab; Drug: Vinblastin

INTERVENTIONS:
Drug: Nivolumab — 240 mg
Drug: Vinblastin — 6mg/m²

SUMMARY:
This study is a multicentric phase II open-label trial consisting of 6 cycles Nivolumab (2 weeks interval) followed by a PET-CT scan. The treatment will be allocated according to PET and CT scan responses. :

* In case of CMR according to Lugano Classification (Cheson et al.2014, PET-CT based response), patients will receive 18 additional cycles of Nivolumab, according to CT-based response at Cycle 12.
* In case of Partial Metabolic Response (PMR) or No Metabolic Response(NMR), according to Lugano Classification (Cheson et al.2014, PET-CT based response) patients will receive 12 to 18 cycles of Nivolumab combined with Vinblastin according to CT-based response at Cycle 12.
* In case of progressive disease, according to Lugano Classification (Cheson et al.2014, PET-CT scan based response) patients will be considered in treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of classical Hodgkin lymphoma according to World Health Organization (WHO) criteria excluding nodular lymphocyte predominant subtype
* Age 61 years or older
* Unfit for poly chemotherapy because of co-morbidities evaluated by a Cumulative Illness Rating Scale (CIRS) score ≥6)
* No previous treatment for Hodgkin lymphoma
* Ann Arbor stages: I-IV
* Baseline 18-fluoro-2-deoxy-D-glucose (18F-FDG) PET-CT (PET0) performed before any treatment with at least one hypermetabolic lesion
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* minimum life expectancy of 3 months
* covered by a social security system
* Men who are sexually active with women with childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug and for at least 7 months after the last drug administration.

Exclusion Criteria:

* Contra-indication to Nivolumab and /or Vinblastin
* Subjects with active interstitial pneumonitis
* Subjects with active infectious disease
* Subjects with active, known or suspected autoimmune disease. Are permitted to enroll: subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Any serious active disease, severe cardio-pulmonary, or metabolic disease interfering with normal application of protocol treatment (according to the investigator's decision)
* Any of the following abnormal laboratory values (unless due to underlying HL) :

  1. Calculated creatinine clearance < 30 mL/min (MDRD formula)
  2. aspartate transaminase (AST) or alanine transaminase (ALT) > 2.5 times the upper limit of normal (ULN)
  3. Serum total bilirubin > 30µmol/L
  4. Neutrophils<1 G/L or Platelets<50 G/L, (unless related to bone infiltration by lymphoma)
* Any history of cancer evolution requiring therapy during the last 3 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma. Patients previously diagnosed with prostate cancer are eligible if :

  1. Their disease was T1-T2a, N0, M0, with a Gleason score ≤ 7, and a prostate specific antigen (PSA) ≤ 10 ng/mL prior to initial therapy,
  2. They had definitive curative therapy (ie, prostatectomy or radiotherapy) ≥ 2 years before Day 1 of Cycle 1,
  3. At a minimum 2 years following therapy they had no clinical evidence of prostate cancer, and their PSA was undetectable if they underwent prostatectomy or <1 ng/mL if they did not undergo prostatectomy.
* Uncontrolled diabetes mellitus leading to impossibility to perform PET scan
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study
* Adult person under legal protection
* Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness
* Subjects with know Human Immunodeficiency Virus (HIV) positivity
* Subjects with known active hepatitis B (HB) infection (positive Ag HB s or positive DNA polymerase chain reaction (PCR) or positive antibody anti-HB c with lack of antibody against HBs) or active hepatitis C infection (patients with positive HCV serology are eligible only if PCR is negative for known hepatitis C virus (HCV RNA)
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Complete Metabolic Response (CMR) rate (Deauville scale 1-3) at the end of treatment | 12 months
  by the Lugano classification 2014

SECONDARY OUTCOMES:
Quantity of drug taken | 12 months
Number of Serious Adverse Event | 12 months
Progression-free survival (PFS) | 5 years
Event-free survival (EFS) | 5 years
Overall survival (OS) | 5 years
Complete Metabolic Response (CMR) rate | 3 months
  by the Lugano classification 2014 at the end of induction treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincent RIBRAG, Study Chair — Institut Gustave Roussy Cancer, Villejuif, France - LYSA; Julien LAZAROVICI, Study Chair — Institut Gustave Roussy Cancer, Villejuif, France - LYSA; Marc ANDRE, Study Chair — CHU Dinant Godinne, UCL Namur, Yvoir - Belgium - LYSA
Locations (51):
- Belgium (9):
  - ZNA Stuivenberg, Antwerp
  - Az Sint Jan, Bruges
  - Clinique Universitaire Saint LUC, Brussels
  - Institut Jules Bordet, Brussels
  - Hopital Jolimont, Haine-Saint-Paul
  - Az Groeninge, Kortrijk
  - CHU de Liege, Liège
  - CHU Dinant Godinne, Yvoir
  - CHU UCL Namur, Yvoir
- France (42):
  - CHU d'Amiens, Amiens
  - CH d'Avignon - Hôpital Henri Duffaut, Avignon
  - CH Côte Basque, Bayonne
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié - Bordeaux, Bordeaux
  - Institut d'Hématologie de Basse Normandie - CHU Côte de Nacre, Caen
  - CH Métropole Savoie, Chambéry
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CH Sud Francilien de Corbeil, Corbeil-Essonnes
  - APHP-Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CHU de Grenoble, Grenoble
  - CHD de Vendée, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH du Mans, Le Mans
  - CH Saint Vincent de Paul, Lille
  - CHRU de LILLE - Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - CHRU de Metz-Thionville, Metz
  - CHU de Montpellier - Saint Eloi, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU de Nîmes - Caremeau, Nîmes
  - APHP - Hopital Necker, Paris
  - APHP - Hôpital de la Pitié Salpetrière, Paris
  - APHP - Hôpital Saint Louis, Paris
  - Centre François Magendie - Hôpital du Haut Lévêque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de La Milétrie, Poitiers
  - Ch Rene Dubos, Pontoise
  - Centre Hospitalier Annecy-Genevois - Site d'Annecy, Pringy
  - CHU Robert Debré, Reims
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - CH de Saint Brieuc, Saint-Brieuc
  - CHRU de Strasbourg, Strasbourg
  - IUCT Toulouse, Toulouse
  - CHU Bretonneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No